CLINICAL TRIAL: NCT03860740
Title: Effect of Physical Exercise on Ki-67 Levels in Women With Operable Breast Cancer Hormonal Receptor Positive, HER2 Negative
Brief Title: Effect of Physical Exercise on Tumor Proliferation of Luminal B Breast Cancer Patients
Acronym: EFIK
Status: Completed | Type: Observational
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other); Faculty of Physical Activity and Sport Sciences (INEF) (Unknown)
Responsible Party: Sponsor
Other Study IDs: GEICAM/2014-09
Record Dates: First submitted 2017-01-13; First posted 2019-03-04 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer; Luminal B
Keywords: Physical exercise; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor samples Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High intensity physical exercise: Supervised Exercise Group: Customized and supervised exercise high intensity training program during 2-3 weeks previous surgery.
  Interventions: Other: Exercise
- Control: Supervised Stretching Group: a stretching and body balance classes will be developed to control the possible confounders and to control the exercise level of participants.
  Interventions: Other: Stretching

INTERVENTIONS:
Other: Exercise — Exercise intervention adapted to maximum rate of oxygen consumption measured during incremental exercise (VO2level) of each patient, working between 60% to 100% VO2level. The activity will be walk-run in a treadmill. 10 sessions minimum
  Groups: High intensity physical exercise
Other: Stretching — Stretching and relaxing exercise during 30 minutes. Same number of sessions as intervention group
  Groups: Control

SUMMARY:
Observational study to evaluate the effect of physical exercise prior to surgery and adjuvant systemic treatment in women with newly diagnosed operable hormone receptor(HR)-positive, human epidermal growth factor receptor 2 (HER2)-negative breast cancers

DETAILED DESCRIPTION:
Effect of exercise on tumor aggressiveness and the impact on patients' quality of life.

Exercise is a safe and effective treatment for women diagnosed with breast cancer (BC), that has an integral benefit during and after treatments, however, the effect at the tumour microenvironment it is unknown; previous studies have evaluated the association between exercise and BC, finding a positive influence on it, which suggest that exercise could reduce the aggressiveness of the tumour. This study will explore the exercise impact in tumor microenvironment, as part of the therapy given to the patients prior to surgery and treatment. In addition, different serum biomarkers involved and the tailoring of exercise for these women will be evaluated. The effect of exercise on treatments secondary effects, biomarkers and quality of life will be evaluated after 6 months of BC surgery. This project will open a window of opportunity to explore new translational research as well as new treatment vias to the patients of this breast cancer subgroup.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, previously untreated clinical stage I-IIIA without previous treatment.
* ER positive breast cancer according to local results. (RH+ is defined as ≥ 1% assessed by Immunohistochemistry (IHC) to Estrogen Receptor (ER) and/or Progesterone Receptor (P)E).
* HER2 negative in the primary tumour according to local results. (HER2 confirmation should be done following the American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) 2013 guidelines)
* Scheduled to undergo surgical resection.
* Ki67 levels must be over 13%, according to local results.
* At least 14 days from enrolment to planned surgical resection.
* Karnofsky performance status of at least 70% at study entry or 0-1 level in Eastern Cooperative Oncology Group (ECOG) Scale.
* Signed consent prior to initiation of study-related procedures.

Exclusion Criteria:

* Schedule to receive any form of induction/neoadjuvant therapy
* Significant cardiac disease (ventricular ejection fraction of <50%, unstable angina, placement of cardiac stents and myocardial infarction within precious 6 months)
* Any pulmonary dysfunction which may affect to the exercise program perform.
* Any mental disease or condition that compromise the physical, psychological and emotional patients' wellness or affect to the process.
* Contraindications to a cardiopulmonary exercise test as recommended by the American Thoracic Society.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with newly diagnosed operable hormone receptor(HR)-positive, human epidermal growth factor receptor 2 (HER2)-negative breast cancers
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
Tumor proliferation (Ki67) | Post-surgery, an average of 6 months
  Tumor proliferation (Ki67) will be assessed immunohistochemically at basal biopsies versus post-surgery tumor samples.
Proliferation Score | Post-surgery, an average of 6 months
  A 50-gene quantitative polymerase chain reaction (qPCR) assay (PAM50) will be used to identify the intrinsic biological subtypes using RNA isolated from formalin-fixed, paraffin-embedded (FFPE) tissue from baseline biopsies samples and post-surgery tumor samples.

SECONDARY OUTCOMES:
Change from baseline molecular subtypes | Post-surgery, an average of 6 months
  A 50-gene qPCR assay (PAM50) will be used to identify the intrinsic biological subtypes using RNA isolated from formalin-fixed, paraffin-embedded (FFPE) tissue from baseline biopsies samples and post-surgery tumor samples.
Changes in tumor microenvironment: levels of Vascular endothelial growth factor (VEGF) | Post-surgery, an average of 6 months
  VEGF will be evaluated on tissue from baseline biopsies samples and post-surgery tumor samples by Immunohistochemistry (IHC)
Changes in tumor microenvironment: levels of factor Hypoxia-inducible factor 1 (HIF-1) | Post-surgery, an average of 6 months
  HIF-1 will be evaluated on tissue from baseline biopsies samples and post-surgery tumor samples by Immunohistochemistry (IHC)
Change in tumor microenvironment: levels of cleaved caspase 3 | Post-surgery, an average of 6 months
  Levels of cleaved caspase 3 will be evaluated on tissue from baseline biopsies samples and post-surgery tumor samples by Immunohistochemistry (IHC)
Oxygen uptake during peak exercise (VO2peak) | Post-surgery, an average of 6 months
  VO2peak will be obtained of the Cardiopulmonary exercise testing (CPET) performed at baseline and after the exercise program until surgery.
Change in body composition | Post-surgery, an average of 6 months
  Change in body composition will be assessed by bioimpedance parameters. Bioelectrical impedance analysis (BIA) is a commonly used method for estimating body composition, and in particular body fat, and will be performed at baseline and after the exercise program until surgery.
Change in fatigue levels | Post-surgery, an average of 6 months
  Change in fatigue levels will be assessed by questionnaire Functional Assessment of Cancer Therapy: Fatigue (FACT-F). The physical well-being domain has 7 items with scores from 0 to 28 points; social/family well-being, 7 items with score from 0 to 28 points; emotional well-being, 6 items with score from 0 to 24 points; functional well-being, 7 items with score from 0 to 28 points; and fatigue subscale, 13 items with score from 0 to 52. Each item has ﬁve likert-type options graduated from 0 to 4: "Not at all", "A little bit"; Somewhat"; "Quite a bit"; "Very much'. The ﬁnal score of FACT-F is obtained by adding the scores of the ﬁve domains, and may vary from 0 to 160 points. The higher the number of points, the better the quality of life and the less the fatigue of the patients is. To obtain the score, the negative questions are reverted; then the answers of the domains are added up, and a proportional average is carried out in case of non answered items.
Change in quality of life levels | Post-surgery, an average of 6 months
  Change in quality of life levels will be assessed by questionnaire Functional Assessment of Cancer Therapy: Breast Cancer (FACT-B). The FACT-B is a breast cancer-specific HRQoL instrument of the FACIT system. The 37-item are divided into five subscales, namely physical (PWB), social/family (SWB), emotional (EWB), functional well-beings (FWB), and the additional concerns for breast cancer (BCS). Each item is rated on a 5-point Likert scale. Negatively worded items were recoded such that a higher score indicates a better HRQoL. The FACT-B total score is the sum of scores of all five subscales.
Change in depression levels | Post-surgery, an average of 6 months
  Change in depression levels will be assessed by questionnaire Center for Epidemiologic Studies Depression Scale (CES-D). The CES-D is a 20-item measure assessing symptoms of depression with items phrased as self-statements (e.g., "I felt hopeful about the future"). Respondents rate how frequently each item applied to them over the course of the past week. Ratings were based on a 4-point Likert scale ranging from 0 (rarely or none of the time [less than 1 day]) to 3 (most or all of the time [5-7 days]).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital General Universitario Gregorio Marañón; Study Director, Study Director — Fundación Jimenez Díaz
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chirlaque MD, Salmeron D, Ardanaz E, Galceran J, Martinez R, Marcos-Gragera R, Sanchez MJ, Mateos A, Torrella A, Capocaccia R, Navarro C. Cancer survival in Spain: estimate for nine major cancers. Ann Oncol. 2010 May;21 Suppl 3:iii21-29. doi: 10.1093/annonc/mdq082. PMID 20427356
- [Background] Bertolini F. Adipose tissue and breast cancer progression: a link between metabolism and cancer. Breast. 2013 Aug;22 Suppl 2:S48-9. doi: 10.1016/j.breast.2013.07.009. PMID 24074792
- [Background] Mishra SI, Scherer RW, Geigle PM, Berlanstein DR, Topaloglu O, Gotay CC, Snyder C. Exercise interventions on health-related quality of life for cancer survivors. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD007566. doi: 10.1002/14651858.CD007566.pub2. PMID 22895961
- [Background] Jones LW, Liang Y, Pituskin EN, Battaglini CL, Scott JM, Hornsby WE, Haykowsky M. Effect of exercise training on peak oxygen consumption in patients with cancer: a meta-analysis. Oncologist. 2011;16(1):112-20. doi: 10.1634/theoncologist.2010-0197. Epub 2011 Jan 6. PMID 21212429
- [Background] Herrero F, San Juan AF, Fleck SJ, Balmer J, Perez M, Canete S, Earnest CP, Foster C, Lucia A. Combined aerobic and resistance training in breast cancer survivors: A randomized, controlled pilot trial. Int J Sports Med. 2006 Jul;27(7):573-80. doi: 10.1055/s-2005-865848. PMID 16802254
- [Background] Jones LW, Demark-Wahnefried W. Diet, exercise, and complementary therapies after primary treatment for cancer. Lancet Oncol. 2006 Dec;7(12):1017-26. doi: 10.1016/S1470-2045(06)70976-7. PMID 17138223
- [Background] Schmitz KH, Ahmed RL, Yee D. Effects of a 9-month strength training intervention on insulin, insulin-like growth factor (IGF)-I, IGF-binding protein (IGFBP)-1, and IGFBP-3 in 30-50-year-old women. Cancer Epidemiol Biomarkers Prev. 2002 Dec;11(12):1597-604. PMID 12496050
- [Background] Battaglini C, Bottaro M, Dennehy C, Rae L, Shields E, Kirk D, Hackney AC. The effects of an individualized exercise intervention on body composition in breast cancer patients undergoing treatment. Sao Paulo Med J. 2007 Jan 4;125(1):22-8. doi: 10.1590/s1516-31802007000100005. PMID 17505681
- [Background] Demark-Wahnefried W, Case LD, Blackwell K, Marcom PK, Kraus W, Aziz N, Snyder DC, Giguere JK, Shaw E. Results of a diet/exercise feasibility trial to prevent adverse body composition change in breast cancer patients on adjuvant chemotherapy. Clin Breast Cancer. 2008 Feb;8(1):70-9. doi: 10.3816/CBC.2008.n.005. PMID 18501061
- [Background] Demark-Wahnefried W, Kenyon AJ, Eberle P, Skye A, Kraus WE. Preventing sarcopenic obesity among breast cancer patients who receive adjuvant chemotherapy: results of a feasibility study. Clin Exerc Physiol. 2002 Feb;4(1):44-49. PMID 16946801
- [Background] Irwin ML, McTiernan A, Baumgartner RN, Baumgartner KB, Bernstein L, Gilliland FD, Ballard-Barbash R. Changes in body fat and weight after a breast cancer diagnosis: influence of demographic, prognostic, and lifestyle factors. J Clin Oncol. 2005 Feb 1;23(4):774-82. doi: 10.1200/JCO.2005.04.036. PMID 15681521
- [Background] Speck RM, Courneya KS, Masse LC, Duval S, Schmitz KH. An update of controlled physical activity trials in cancer survivors: a systematic review and meta-analysis. J Cancer Surviv. 2010 Jun;4(2):87-100. doi: 10.1007/s11764-009-0110-5. Epub 2010 Jan 6. PMID 20052559
- [Background] Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvao DA, Pinto BM, Irwin ML, Wolin KY, Segal RJ, Lucia A, Schneider CM, von Gruenigen VE, Schwartz AL; American College of Sports Medicine. American College of Sports Medicine roundtable on exercise guidelines for cancer survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409-26. doi: 10.1249/MSS.0b013e3181e0c112. PMID 20559064
- [Background] Ibrahim EM, Al-Homaidh A. Physical activity and survival after breast cancer diagnosis: meta-analysis of published studies. Med Oncol. 2011 Sep;28(3):753-65. doi: 10.1007/s12032-010-9536-x. Epub 2010 Apr 22. PMID 20411366
- [Background] Irwin ML. Physical activity interventions for cancer survivors. Br J Sports Med. 2009 Jan;43(1):32-8. doi: 10.1136/bjsm.2008.053843. Epub 2008 Oct 23. PMID 18948351
- [Background] Betof AS, Dewhirst MW, Jones LW. Effects and potential mechanisms of exercise training on cancer progression: a translational perspective. Brain Behav Immun. 2013 Mar;30 Suppl(0):S75-87. doi: 10.1016/j.bbi.2012.05.001. Epub 2012 May 17. PMID 22610066
- [Background] Holmes MD, Chen WY, Feskanich D, Kroenke CH, Colditz GA. Physical activity and survival after breast cancer diagnosis. JAMA. 2005 May 25;293(20):2479-86. doi: 10.1001/jama.293.20.2479. PMID 15914748
- [Background] Jones LW, Peddle CJ, Eves ND, Haykowsky MJ, Courneya KS, Mackey JR, Joy AA, Kumar V, Winton TW, Reiman T. Effects of presurgical exercise training on cardiorespiratory fitness among patients undergoing thoracic surgery for malignant lung lesions. Cancer. 2007 Aug 1;110(3):590-8. doi: 10.1002/cncr.22830. PMID 17582629
- [Background] Burgomaster KA, Hughes SC, Heigenhauser GJ, Bradwell SN, Gibala MJ. Six sessions of sprint interval training increases muscle oxidative potential and cycle endurance capacity in humans. J Appl Physiol (1985). 2005 Jun;98(6):1985-90. doi: 10.1152/japplphysiol.01095.2004. Epub 2005 Feb 10. PMID 15705728
- [Background] Rao R, Cruz V, Peng Y, Harker-Murray A, Haley BB, Zhao H, Xie XJ, Euhus D. Bootcamp during neoadjuvant chemotherapy for breast cancer: a randomized pilot trial. Breast Cancer (Auckl). 2012;6:39-46. doi: 10.4137/BCBCR.S9221. Epub 2012 Feb 1. PMID 22399859
- [Background] Jones LW, Fels DR, West M, Allen JD, Broadwater G, Barry WT, Wilke LG, Masko E, Douglas PS, Dash RC, Povsic TJ, Peppercorn J, Marcom PK, Blackwell KL, Kimmick G, Turkington TG, Dewhirst MW. Modulation of circulating angiogenic factors and tumor biology by aerobic training in breast cancer patients receiving neoadjuvant chemotherapy. Cancer Prev Res (Phila). 2013 Sep;6(9):925-37. doi: 10.1158/1940-6207.CAPR-12-0416. Epub 2013 Jul 10. PMID 23842792
- [Background] Pedersen BK. Muscle as a secretory organ. Compr Physiol. 2013 Jul;3(3):1337-62. doi: 10.1002/cphy.c120033. PMID 23897689
- [Background] Jones LW, Viglianti BL, Tashjian JA, Kothadia SM, Keir ST, Freedland SJ, Potter MQ, Moon EJ, Schroeder T, Herndon JE 2nd, Dewhirst MW. Effect of aerobic exercise on tumor physiology in an animal model of human breast cancer. J Appl Physiol (1985). 2010 Feb;108(2):343-8. doi: 10.1152/japplphysiol.00424.2009. Epub 2009 Dec 3. PMID 19959769
- [Background] Irwin ML, Smith AW, McTiernan A, Ballard-Barbash R, Cronin K, Gilliland FD, Baumgartner RN, Baumgartner KB, Bernstein L. Influence of pre- and postdiagnosis physical activity on mortality in breast cancer survivors: the health, eating, activity, and lifestyle study. J Clin Oncol. 2008 Aug 20;26(24):3958-64. doi: 10.1200/JCO.2007.15.9822. PMID 18711185
- [Background] Zeng H, Irwin ML, Lu L, Risch H, Mayne S, Mu L, Deng Q, Scarampi L, Mitidieri M, Katsaros D, Yu H. Physical activity and breast cancer survival: an epigenetic link through reduced methylation of a tumor suppressor gene L3MBTL1. Breast Cancer Res Treat. 2012 May;133(1):127-35. doi: 10.1007/s10549-011-1716-7. Epub 2011 Aug 12. PMID 21837478
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org